CLINICAL TRIAL: NCT01157520
Title: Hypotensive Episodes During Cesarean Section Detected by a Continuous Non-invasive Arterial Pressure Measurement Device Are Missed by the Oscillometric Blood Pressure Measurement
Brief Title: Study to Detect Hypotensive Episodes During Spinal Anesthesia for Cesarean Section Using a Noninvasive Continuous Device
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Other Study IDs: CNAP_Sectio
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cesarean: Women scheduled for elective Cesarean section under spinal anesthesia

SUMMARY:
Hypotension after spinal anesthesia for Cesarean section occurs in up to 90% usually under five minutes after local anesthetics administration. These changes are poorly depicted by oscillometric measurements. The investigators hypothesized, that a continuous noninvasive device detects more hypotensive periods with lower blood pressures.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* week of pregnancy >36

Exclusion Criteria:

* emergency cases

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: elective Cesarean section under spinal anesthesia
Sampling Method: Probability Sample
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)